CLINICAL TRIAL: NCT06898619
Title: The Impact of Crisis Management Training on Disaster Nursing Competencies: a Pre-Test and Post-Test Evaluation
Brief Title: The Impact of Crisis Management Training on Disaster Nursing Competencies
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Seda Tugba Baykara Mat, Asst. Prof., University of Beykent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Crisis management
Record Dates: First submitted 2025-01-21; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-01

CONDITIONS: Crisis Intervention
Keywords: Crisis Management; Disaster Nursing; Pretest-Posttest Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nursing students 3. grade (Experimental): To equip third-year nursing students with the necessary knowledge, skills, and strategies to effectively manage crises in healthcare settings, ensuring patient safety and optimal care delivery.
  Interventions: Behavioral: Crisis Management Training for Third-Year Nursing Students

INTERVENTIONS:
Behavioral: Crisis Management Training for Third-Year Nursing Students — Crisis management is essential for nurses, who often work on the front lines during emergencies. This training program for third-year nursing students equips them with the skills and knowledge required to handle crises effectively. The program includes nine stages: raising awareness, assessing baseline knowledge, reinforcing foundational concepts, introducing advanced techniques, practicing through simulations, reflecting on learning, providing feedback, summarizing key points, and enhancing learning with additional resources.
  Participants explore critical topics such as disaster response, triage, communication strategies, and teamwork. Simulated scenarios help develop practical skills like decision-making and prioritization under pressure. Feedback and reflective discussions reinforce learning, while additional resources encourage ongoing professional growth.
  By bridging theoretical knowledge with practical application, the training prepares nursing students to respond confidently t

SUMMARY:
This study aims to evaluate the effectiveness of crisis management training designed for third-year nursing students. Crisis management in the healthcare sector holds critical importance during unforeseen events such as natural disasters and emergencies. The ability of nurses to effectively plan, make quick decisions, and manage crises successfully plays a vital role in ensuring patient safety and operational efficiency. The primary objective of this research is to enhance nursing students' crisis management skills and to assess the extent to which these skills can be improved through targeted training.

The study employs a pre-test and post-test design. The participants will consist of third-year nursing students. A pre-test will be administered before the training to assess the participants' existing knowledge and skills in crisis management. The training content will focus on crisis management concepts, planning strategies, rapid decision-making processes, and team coordination. Additionally, intervention approaches to natural disasters such as earthquakes will be addressed in detail. At the conclusion of the training, a post-test will be conducted to evaluate the program's effectiveness.

The data collection process will utilize the Disaster Nursing Preparedness and Response Competency Scale, a standardized tool designed to measure students' levels of preparedness, problem-solving skills during crises, and intervention effectiveness. The training program will adopt an interactive approach, integrating both theoretical and practical components.

The study hypothesizes that crisis management training will significantly enhance the disaster nursing competencies of nursing students. The findings aim to reveal whether the training leads to a substantial improvement in the knowledge and skill levels of the participants.

The study is scheduled to be conducted at a private university in Istanbul in March 2025. The study population comprises all third-year nursing students enrolled in the nursing program at the university during the study period (N=70). No sampling method will be used, as the study aims to include the entire population. The training program will consist of a single session and will incorporate feedback from students and motivation-enhancing activities. Slavin's Effective Teaching Model will be employed, featuring presentations and interactive sessions. Data will be collected using a Personal Information Form and the Disaster Nursing Preparedness and Response Competency Scale.

The collected data will be analyzed using SPSS for Windows 22.0. The normality of data distribution will be assessed using the Kolmogorov-Smirnov Test. If the Kolmogorov-Smirnov Test indicates p>0.05p > 0.05p>0.05, the data will be considered normally distributed. Conversely, if p<0.05p < 0.05p<0.05, the data will be deemed non-normally distributed, and skewness and kurtosis values will be examined. Changes in repeated measurements will be analyzed using a Repeated Measures ANOVA if the data is normally distributed, or the Friedman Test if it is not.

Descriptive statistics will be employed to summarize the general characteristics of the data, including the means and distributions of pre-test and post-test scores. To evaluate the impact of the training program, a Paired Samples T-Test will be conducted to assess the differences between pre-test and post-test scores within the same group. This analysis will measure the program's effects on time management and procrastination behaviors. Additionally, effect sizes (e.g., Cohen's d) will be calculated to evaluate the magnitude and significance of the intervention's effects.

Variance analysis (ANOVA) may also be used to determine significant differences between groups if deemed necessary. Furthermore, a Power Analysis will be conducted to assess whether the study has an adequate sample size. These analyses will provide meaningful and reliable interpretations of the study findings.

ELIGIBILITY:
Inclusion Criteria:

* Must be over 18 years of age.
* Must be enrolled as a third-year nursing student at the university where the research is conducted.
* Must be attending full-time education.
* Must have a sufficient level of proficiency in Turkish to understand and communicate.
* Must voluntarily agree to participate.

Exclusion Criteria:

* Change of department/school
* Request by the student to withdraw from the study
* Being under 18 years of age
* Inability to understand Turkish at a sufficient level

Min Age: 18 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-25 (Estimated)

PRIMARY OUTCOMES:
Disaster Nursing Preparedness and Response Competency | 3 weeks
  In the study, a 34-item scale was used. The correlation coefficients between the total score of the scale and the item scores, as well as the correlation coefficients between the subscale scores and the total score, were found to be positively high, distinctive, and reliable. In confirmatory factor analysis, the fit indices and factor loadings were appropriate, and the two-section, seven-subscale structure of the scale was found to be valid. The Cronbach's Alpha coefficient was calculated to be between 0.89 and 0.95 for the subscales, 0.95 for the sections, and 0.97 for the entire scale, indicating high internal consistency. The correlation between the equivalent halves analysis was found to be 0.97, and the Spearman-Brown coefficient calculated using this correlation was determined to be 0.98. In the Guttman split-half analysis, all Lambda coefficients were higher than 0.9. Based on these results, the scale's reliability in terms of internal consistency was confirmed.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Beykent University, Istanbul, Beylikduzu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No